CLINICAL TRIAL: NCT05574140
Title: BreathinG-induced Myocardial and Cerebral Perfusion in Anxiety Disorders (B-GLAD)
Brief Title: BreathinG-induced Myocardial and Cerebral Perfusion in Anxiety Disorders
Acronym: B-GLAD
Status: Recruiting | Type: Observational
Sponsor: McGill University Health Centre/Research Institute of the McGill University Health Centre (Other)
Responsible Party: Principal Investigator, Matthias Friedrich, Principal Investigator, McGill University Health Centre/Research Institute of the McGill University Health Centre
Other Study IDs: 2020-6298
Record Dates: First submitted 2022-10-06; First posted 2022-10-10 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-04

CONDITIONS: Generalized Anxiety Disorder; Oxygenation Sensitive CMR
MeSH Terms: conditions — Generalized Anxiety Disorder

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patient Population: Participants diagnosed with Generalized Anxiety Disorder
  Interventions: Diagnostic Test: Cardiac MRI
- Healthy Volunteers: Participants with no pre-existing conditions and who are on no medications.
  Interventions: Diagnostic Test: Cardiac MRI

INTERVENTIONS:
Diagnostic Test: Cardiac MRI — The 4-minute breathing maneuver comprised of 2 minutes of normal breathing and 1-min hyperventilation (rate of 30 breaths per minute) followed by a maximal breath-hold. This technique is used in Oxygenation Sensitive CMR, a type of MRI, and will induce a vasoactive response visible in cardiac and cerebral MRI images
  Other Names: Breathing Maneuvers

SUMMARY:
This study aims to view variations in MRI measurements of the heart and the brain in people with anxiety versus healthy volunteers. The MRI measurements used will be Oxygenation-Sensitive Cardiac MRI (OS-CMR), a recent type of MRI which is safe, fast, and non-invasive.

DETAILED DESCRIPTION:
The investigators will prospectively analyze OS-CMR data from patients with a generalized anxiety disorder from one site. The investigators will observe how an anxiety disorder affects the OS-CMR data. In a follow-up MRI scan, the investigators will look at the OS-CMR of a subgroup who have anxiety disorder and are also undertaking cognitive behavioural therapy to asses how and if this therapy affects the OS-CMR data.

ELIGIBILITY:
Inclusion Criteria:

Patient population:

Age 18-55,

* Confirmation of an anxiety disorder as identified by the PSWQ,
* No known, current or history, of significant medical conditions that may affect or directly involve the neurological, cardiovascular or respiratory system (except anxiety and depression)
* Non-smoker

Healthy Volunteers:

* Age 18-55
* No known, current or history, of significant medical conditions that may affect or directly involve the neurological, cardiovascular or respiratory system
* Non-smoker

Exclusion Criteria:

* General MRI contraindications: pacemakers, defibrillating wires, implanted defibrillators, intracranial aneurysm clips, metallic foreign bodies in the eyes, pregnancy
* History of significant neurological disease or illness that is not anxiety (e.g. Dementia, stroke)
* Hemodynamically unstable conditions
* Significant or uncontrolled arrhythmias
* Severe pulmonary disease
* Recent (<90 days) myocardial infarction
* Recent (<90 days) surgery or coronary intervention
* Consumption of caffeine (caffeinated beverages, coffee, tea, cocoa, chocolate) within 12h of the exam
* Use of benzodiazepines or other short-acting anxiety medications (<1 day)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study will recruit patient participants who are identified as having Generalized Anxiety Disorder (GAD), as well as age-similar healthy volunteer participants.
Sampling Method: Non-Probability Sample
Enrollment: 84 (Estimated)
Dates: Start 2022-07-15 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
Change in Signal Intensity | Baseline
  Change in signal intensity between the baseline signal intensity and the signal intensity at 30 seconds of breath hold

CONTACTS AND LOCATIONS:
Locations (1):
- Emotional Health CBT Clinic, Montreal, Quebec, Canada